## COMPLUTENSE UNIVERSITY OF MADRID FACULTY OF NURSING, PHYSIOTHERAPY AND PODIATRY



## TITLE:

# CLINICAL TRIAL WITHOUT MEDICATION: PREVENTION OF BODY IMAGE DISORDER FOR NURSING INTERVENTION ON PATIENT AND FAMILY PRIOR TO MAMA AND COLON CANCER SURGERY

## MEMORY TO CHOOSE THE DEGREE OF DOCTOR PRESENTED BY

Natalia Mudarra García

Under the direction of the doctors

Enrique Pacheco Del Cerro Alfonso Meneses Morroy

Madrid, 2018

#### PROCEDURE FOR ANALYSIS AND INTERPRETATION OF DATA:

The data collection lasted one and a half years, from April 2017 to August 2018. Once collected, they were coded in a database and later analyzed through the statistical program SPSS 21.

All the study variables were analyzed descriptively, in order to study the distribution of the same. The categorical variables were described by the associated percentage for each of the possible response options, and the quantitative variables by means of the mean, the standard deviation and the range.

To verify the normality of the data, the Kolmogorov-Smirnov test was used for a sample with quantitative variables. This test indicates whether our sample has a normal distribution (p> 0.05) or, on the contrary, it is not distributed normally (p $\leq$ 0.05). For this we have calculated the distribution of each quantitative variable in each group (control and study).

For the contrast of hypothesis and comparisons between the variables of body image, self-esteem and quality of life were used: the Chi square test for categorical variables, the Student's t test or ANOVA for quantitative variables that are distributed in a normal way, and the Mann-Whitney U test or Kruskal-Wallis test for quantitative variables that do not follow a normal distribution.

To identify the variables that influenced the dependent variable, the Pearson Correlation Coefficient was used. With this index, the joint correlation between the dependent variable (body image disorder) and the independent variables (study group, body image, self-esteem and quality of life) was measured.

A linear regression model was developed to determine the effect of the dependent variable (body image disorder) on the independent variable (go with or without a relative).

### **RESULTS**

The subjects who underwent breast surgery were 188 patients and those who underwent colorectal surgery were 15 in total.

Of the 188 patients who were going to undergo breast surgery, 136 were excluded because they did not meet the inclusion criteria: 31 were excluded because they had received neoadjuvant therapy, 91 because they were benign, 5 had been operated on previously, 2 rejected the surgery, 2 were male, 3 decided to undergo surgery in another hospital and 2 could not give their consent when being supervised. No patient left the study.

Of the 15 patients who underwent surgery for colon surgery, 3 were excluded because they did not perform a stoma during the surgical procedure.

Finally, 52 patients diagnosed with breast cancer (18 with mastectomy and 34 with conservative surgery) and 12 patients diagnosed with colorectal cancer with ostomy participated in the study.

| | | Control | Study | Total | P |
|---|---|---|---|---|---|
| | | N=32 | N=32 | N=64 | |
| | High self-esteem | 28 (87,5%) | 27 (84,4%) | 55 (85,9%) | |
| SELF ESTEEM | Average self-esteem | 3 (9,4%) | 3 (9,4%) | 6 (9,4%) | |
| N (%) | Low self-esteem | 1 (3,1%) | 2 (6,3%) | 3 (4,7%) | 0,839 |

| | Control | Stydy | Total | P |
|---------------------------|------------|------------|------------|--------|
| | N=32 | N=32 | N=64 | |
| BODY IMAGE | 9,66 (5,7) | 1,31 (1,8) | 5,48 (5,9) | <0,001 |
| Mean (standard deviation) | | | | |

| Control | Study | Total | P |
|---------|-------|-------|---|

| | | N=52 | N=52 | N=52 | |
|---|---|---|---|---|---|
| IMPACT OF THE DISEASE: QRQ BR- | Concern for the future | 65,3 (23,5) | 66,3 (26,4) | 65,8 (24,7) | 0,954 |
| 23 | Tutuic | | | | |
| | Sex practice | 29,1 (25,7) | 29,8 (26,5) | 29,5 (25,8) | 0,925 |
| Mean (standard deviation) | Enjoy sex | 29,1 (38) | 27,2 (29,7) | 28,2 (33,9) | 0,700 |
| | Symptomatology of the breast | 50,9 (14,2) | 47,8 (15,2) | 49,3 (14,6) | 0,448 |
| | Symptomatology of the arm | 38,7 (13,3) | 32,9 (14) | 35,8 (13,8) | 0,035 |
| | Symptomatology of the arm | 42,5 (16,3) | 44,4 (19) | 43,4 (17,2) | 0,931 |

| | self esteem | future | PRACTICE<br>OF SEX | ENJOY<br>SEX | SYMPTOMS<br>MAMA | SYMPT<br>OMS<br>ARM |
|---|---|---|---|---|---|---|
| DISORDER OF<br>THE BODY<br>IMAGE | p=0.142 | p=0,828 | p=0,161 | p=0,034 | p=0,137 | p=0,007 |

In the self-esteem perceived by the patient, no statistically significant differences were found between the two groups (p = 0.83).

In the self-esteem perceived by mastectomized women, those undergoing conservative surgery and patients who underwent a stoma, no significant differences were obtained between both groups (p = 0.30) (p = 0.83) (p = 0.29) respectively.

On the other hand, statistically significant differences were obtained in the body image variable between the two groups. (p <0.001). Similarly, separating the groups by type of intervention, mastectomy (p <0.001), conservative surgery (p

<0.001) and ostomy (p = 0.002), statistically significant differences were also obtained in relation to the body image between the control group and the control group. study group.

When analyzing the concern for the future (p = 0.95), sexual activity (p = 0.925) and sex enjoyment (p = 0.70) no statistically significant differences were found between the two groups.

There were no statistically significant differences between the study group and the control group with respect to the symptoms of the breast (p = 0.44).

Statistically significant results were obtained in the arm symptomatology (p = 0.035) between both groups.

Analyzing only the patients undergoing mastectomy, no statistically significant differences were obtained in relation to the worry about the future (p = 0.954), sex practice (p = 0.925), sex enjoyment (p = 0.700), breast symptomatology (p = 0.448) and arm (p = 0.035) between both groups.

Selecting only the patients undergoing conservative surgery, no statistically significant differences were found in the variables concern for the future (p = 0.946), sex practice (p = 0.594), enjoyment of sex (p = 0.477) and symptomatology of the breast (p = 0.193), but they were found in the arm symptomatology (p = 0.009) between both groups.

The differences were not statistically significant between body image and self-esteem (p = 0.142), concern for the future (p = 0.828), sex practice (p = 0.161) and breast symptomatology (p = 0.137). On the contrary, if statistically significant results were obtained between body image and enjoyment of sex (p = 0.034) and arm symptomatology (p = 0.007).

## **LINEAR REGRESSION:**

The results show that the fact that the patient, together with his relative, comes to the nursing intervention prior to surgery, generates a reduction of 8.34 points in the scale of the body image disorder.